CLINICAL TRIAL: NCT02644252
Title: Tocotrienol as a Nutritional Supplement in Patients With Advanced Non-small Cell Lung Cancer (NSCLC)
Brief Title: Tocotrienol as a Nutritional Supplement in Patients With Advanced Lung Cancer
Acronym: Toco-Pulm
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The trial was ended prematurely because of a poor accrual rate
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Toco-Pulm
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Vinorelbine; Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Performance status 0-1, Arm A (Experimental): Day 1: Cisplatin 75 mg/m2 plus vinorelbine 25 mg/m2. Day 8: Capsule vinorelbine 50 mg/m2. Tocotrienol 300 mg x 3 daily until progression.
  Interventions: Drug: Day 1: Cisplatin 75 mg/m2; Drug: Day 1: Vinorelbine 25 mg/m2; Drug: Day 8: Capsule vinorelbine 50 mg/m2; Dietary Supplement: Tocotrienol 300 mg x 3 daily until progression
- Performance status 0-1, Arm B (Experimental): Day 1: Cisplatin 75 mg/m2 plus vinorelbine 25 mg/m2. Day 8: Capsule vinorelbine 50 mg/m2. Placebo 1 capsule x 3 daily until progression.
  Interventions: Drug: Day 1: Cisplatin 75 mg/m2; Drug: Day 1: Vinorelbine 25 mg/m2; Drug: Day 8: Capsule vinorelbine 50 mg/m2; Drug: Placebo 1 capsule x 3 daily until progression
- Performance status 2, Arm A (Experimental): Day 1: Carboplatin area under the curve (AUC)=5 plus vinorelbine 30mg/m2. Day 8: Capsule vinorelbine 60 mg/m2. Tocotrienol 300 mg x 3 daily until progression
  Interventions: Drug: Day 1: Carboplatin AUC=5; Drug: Day 1: Vinorelbine 30 mg/m2; Drug: Day 8: Capsule vinorelbine 60 mg/m2; Dietary Supplement: Tocotrienol 300 mg x 3 daily until progression
- Performance status 2, Arm B (Experimental): Day 1: Carboplatin area under the curve (AUC)=5 plus vinorelbine 30mg/m2. Day 8: Capsule vinorelbine 60 mg/m2. Placebo 1 capsule x 3 daily until progression
  Interventions: Drug: Day 1: Carboplatin AUC=5; Drug: Day 1: Vinorelbine 30 mg/m2; Drug: Day 8: Capsule vinorelbine 60 mg/m2; Drug: Placebo 1 capsule x 3 daily until progression

INTERVENTIONS:
Drug: Day 1: Cisplatin 75 mg/m2
  Arms: Performance status 0-1, Arm A; Performance status 0-1, Arm B
Drug: Day 1: Vinorelbine 25 mg/m2
  Arms: Performance status 0-1, Arm A; Performance status 0-1, Arm B
Drug: Day 8: Capsule vinorelbine 50 mg/m2
  Arms: Performance status 0-1, Arm A; Performance status 0-1, Arm B
Drug: Day 1: Carboplatin AUC=5
  Arms: Performance status 2, Arm A; Performance status 2, Arm B
Drug: Day 1: Vinorelbine 30 mg/m2
  Arms: Performance status 2, Arm A; Performance status 2, Arm B
Drug: Day 8: Capsule vinorelbine 60 mg/m2
  Arms: Performance status 2, Arm A; Performance status 2, Arm B
Dietary Supplement: Tocotrienol 300 mg x 3 daily until progression
  Arms: Performance status 0-1, Arm A; Performance status 2, Arm A
Drug: Placebo 1 capsule x 3 daily until progression
  Arms: Performance status 0-1, Arm B; Performance status 2, Arm B

SUMMARY:
There is a need for improving the effect of first-line chemotherapy for lung cancer patients, preferably by using an approach with none or very few side effects.

In this trial the investigators incorporate δ-tocotrienol/placebo as a nutritional supplement on top of standard chemotherapy for patients with advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer, including squamous cell carcinomas, adenocarcinomas and non-neuroendocrine large cell carcinomas
* Patients with advanced stages of NSCLC who are candidates to first-line platinum-based doublet chemotherapy
* Measurable disease by RECIST 1.1
* Age ≥ 18 years.
* Performance status 0-2.
* Adequate bone marrow function, liver function, and renal function (within 7 days prior to inclusion):

  * White blood cells (WBC) ≥ 3.0 * 10^9/l or neutrophils (ANC) ≥ 1.5 * 10^9/l
  * Platelet count ≥ 100 * 10^9/l
  * Hemoglobin ≥ 6 mmol/l
  * Serum bilirubin < 2.0 * upper level of normal (ULN)
  * Serum transaminase ≤ 2.5 * ULN
  * Serum creatinine ≤ 1.5 ULN
* Written and orally informed consent.

Exclusion Criteria:

* Other malignant diseases within 5 years prior to inclusion in the study, except curatively treated basal cell or squamous cell carcinoma of the skin and other types of cancer with minimal risk of recurrence.
* Other experimental therapy or participation in another clinical trial within 28 days prior to treatment initiation.
* Patients who have received prior chemotherapy for NSCLC
* Patients with NSCLC who are candidates to neoadjuvant chemotherapy or curative chemoradiotherapy
* Underlying disease not adequately treated (diabetes, cardiac disease)
* Allergy to the active substance or any of the auxiliary agents
* Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival | From date of randomization until date of first documented progression; assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Christa H Nyhus, MD, Study Chair — Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark